CLINICAL TRIAL: NCT01078389
Title: A Multicenter, Randomized, Double-Blind, Phase 2 Study to Evaluate the Effect of Febuxostat Versus Placebo in Joint Damage in Hyperuricemic Subjects With Early Gout
Brief Title: Effect of Febuxostat on Joint Damage in Hyperuricemic Subjects With Early Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMX-67_204; U1111-1113-8098 (Registry Identifier: WHO)
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Joint Damage
Keywords: Gout; Hyperuricemia; Uric Acid; Drug Therapy
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Febuxostat 40 mg or 80 mg (Experimental): Febuxostat 40 mg or 80 mg (based on serum urate levels at Day 14), capsules, orally, once daily for up to 24 Months.
  Interventions: Drug: Febuxostat
- Placebo (Placebo Comparator): Febuxostat placebo-matching capsules, orally, once daily for up to 24 Months.
  Interventions: Drug: Placebo for Febuxostat

INTERVENTIONS:
Drug: Febuxostat — Febuxostat capsules
  Other Names: Uloric; TMX-67
  Arms: Febuxostat 40 mg or 80 mg
Drug: Placebo for Febuxostat — Febuxostat placebo-matching capsules
  Arms: Placebo

SUMMARY:
This purpose of this study is to assess the effect of febuxostat, once daily (QD), on joint damage in patients with elevated serum urate levels and gout.

DETAILED DESCRIPTION:
Gout is caused by high levels of uric acid in the body, and is associated with a broad range of comorbidities including heart disease, chronic kidney disease and additional risk factors like obesity and high blood pressure. Hyperuricemia, which is defined as an elevation in serum urate levels, develops into gout when urate crystals form from supersaturated body fluids and settle in joints and other organs. Urate-lowering therapy is used to treat hyperuricemia in patients with gout.

Current treatments focus on initiating urate-lowering therapy in hyperuricemic gout patients who have experienced multiple acute gout flares within the past year. However, joint damage caused by crystal deposition may occur much earlier than previously considered. Monosodium urate crystals have been found present in the joints of people with hyperuricemia who do not have any symptoms. The presence of monosodium urate crystals would indicate that after the crystals form, they stay within the joint if serum urate levels are not reduced. Lowering uric acid levels and maintaining them may reduce acute gout flare episodes and possibly halt or reduce joint damage in patients with gout.

This study will evaluate the effect of febuxostat on joint damage in hyperuricemic patients with early gout. All patients will receive gout flare prophylaxis for the first 6 months of the study. Gout flares may also be treated throughout the study.

A variety of imaging techniques are in use to evaluate gout. Plain radiographs (x-rays), Magnetic Resonance Imaging (MRI) and Dual Energy Computed Tomography (DECT) will be utilized in this study. The modified Sharp/Van Der Heijde scoring method (named after Drs. Sharp and Van Der Heijde) for assessment of x-rays has been validated in patients with chronic gout and will be used in this study for evaluating erosion and joint space narrowing. Participants are expected to have 15 visits which will include plain radiographic examinations at 5 visits, 3 Magnetic Resonance Imaging (MRI) examinations and 3 DECT procedures at selected sites.

ELIGIBILITY:
Inclusion Criteria:

* The participant, or the participant's legally acceptable representative, signs a written informed consent form/Health Insurance Portability & Accountability Act (HIPAA) Authorization prior to the initiation of any study procedures.
* Must have a history or presence of gout defined as having one or more of the following conditions of the American Rheumatism Association (ARA) preliminary criteria for the diagnosis of gout

  * A tophus proven to contain urate crystals by chemical or polarized light microscopic means and/or
  * Characteristic urate crystals in the joint fluid and/or
  * History of at least 6 of the following clinical, laboratory and x-ray phenomena*: *More than one flare criteria will be excluded for the purpose of this study if the participant has a history of only a single acute gout flare.

    * More than one attack of acute arthritis*
    * maximum inflammation developed within 1 day
    * monoarticular arthritis
    * redness observed over joints
    * first metatarsophalangeal joint painful or swollen
    * unilateral first metatarsophalangeal joint attack
    * unilateral tarsal joint attack
    * tophus (proven or suspected)
    * hyperuricemia
    * asymmetric swelling within a joint on x-ray
    * sub-cortical cysts without erosions on x-ray
    * joint fluid culture negative for organisms during attacks
  * *More than one flare criteria will be excluded for the purpose of this study if the participant has a history of only a single acute gout flare.
* Is male and at least 18 years of age OR;

  * Female ≥45 years of age and at least 2 years post-menopausal AND has a Follicle Stimulating Hormone (FSH) level ≥40 IU/L OR
  * Female receiving hormone replacement therapy (HRT) must be ≥55 years of age (FSH level not required).
* Has hyperuricemia defined as serum Uric Acid (sUA) level ≥7.0 mg/dL at Screening.
* Has a history of ≤2 (1 or 2) flares. In participants with a history of 2 flares, must have had only one flare in any 12 month period. The primary affected joint will be based on the location of the first gout flare which must be located within right or left metatarsophalangeal (MTP), interphalangeal (IP), ankle, metacarpophalangeal (MCP), Proximal Inter-Phalangeal (PIP), or distal inter-phalangeal (DIP) joints prior to Screening.
* Is capable of understanding and complying with protocol requirements, including scheduled clinic procedures.

Exclusion Criteria:

* Previously on urate-lowering therapy (allopurinol, febuxostat or probenecid).
* Has secondary hyperuricemia (eg due to myeloproliferative disorder or organ transplant).
* Has a history of xanthinuria.
* Has a known hypersensitivity to any component of the febuxostat formulation.
* Has rheumatoid arthritis.
* Has active peptic ulcer disease.
* Has a history of cancer, except basal cell carcinoma of the skin, which has not been in remission for at least 5 years prior to the first dose of study medication.
* Has experienced either a myocardial infarction (MI) or stroke within 90 days prior to the Screening visit.
* Has alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) values greater than 2.0 the upper limit of normal during the Screening period.
* Has a significant medical condition and/or conditions that would interfere with the treatment, safety or compliance with the protocol at the discretion of the Investigator.
* Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse with 5 years prior to the Screening visit. Participant consumes >14 alcoholic beverages/week.
* Has received any investigational medicinal product within 30 days prior to the Screening visit. In addition, the participant has been previously randomized into this study and received at least one dose of double blind study drug treatment.
* Has an estimated Glomerular filtration rate (eGFR) <60 mL/min calculated using the Modification of Diet in Renal Disease (MDRD) formula by the Central Laboratory.
* Has a serum creatinine at Screening greater than 2.0 mg/dL.
* Has a known history of infection with hepatitis B, hepatitis C or human immunodeficiency virus.
* Is a study site employee, or is an immediate family member (ie, spouse, parent, child, and sibling) of a study site employee involved in conduct of this study.
* Is unable to understand verbal or written English or any other language for which a certified translation of the approved informed consent form is available.
* Is required to take excluded medications.
* Magnetic Resolution Imaging:

  * Has a known hypersensitivity to gadolinium
  * Has history of severe asthma
  * Has an electronically, magnetically or mechanically activated implanted device
  * Has any object that could present a potential hazard or interfere with MRI interpretation secondary to the artifact (i.e. metallic foreign bodies)
  * Has a significant medical condition considered by the Investigator (or radiologist) to interfere with the participant's ability to receive gadolinium (eg Sickle cell anemia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2010-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (56):
- United States (56):
  - Mesa, Arizona
  - Tucson, Arizona
  - Burbank, California
  - Carmichael, California
  - Costa Mesa, California
  - Irvine, California
  - Orange, California
  - Rancho Cucamonga, California
  - San Diego, California
  - San Luis Obispo, California
  - Trumbull, Connecticut
  - Boynton Beach, Florida
  - Daytona Beach, Florida
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Sanford, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Honolulu, Hawaii
  - Arlington Heights, Illinois
  - Avon, Indiana
  - Greenfield, Indiana
  - Wichita, Kansas
  - Rockport, Maine
  - Chaska, Minnesota
  - Belzoni, Mississippi
  - Olive Branch, Mississippi
  - Billings, Montana
  - Missoula, Montana
  - Bellevue, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Charlotte, North Carolina
  - Lenoir, North Carolina
  - Shelby, North Carolina
  - Dayton, Ohio
  - Franklin, Ohio
  - Willoughby Hills, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Duncansville, Pennsylvania
  - East Providence, Rhode Island
  - Columbia, South Carolina
  - Rapid City, South Dakota
  - Kingsport, Tennessee
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Southlake, Texas
  - Sugar Land, Texas
  - Arlington, Virginia
  - Burke, Virginia
  - Manassas, Virginia
  - Kenosha, Wisconsin

REFERENCES:
- [Derived] Dalbeth N, Saag KG, Palmer WE, Choi HK, Hunt B, MacDonald PA, Thienel U, Gunawardhana L. Effects of Febuxostat in Early Gout: A Randomized, Double-Blind, Placebo-Controlled Study. Arthritis Rheumatol. 2017 Dec;69(12):2386-2395. doi: 10.1002/art.40233. PMID 28975718
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 65 investigative sites in the United States from 10 March 2010 to 3 September 2013.
Pre-assignment Details: Participants with a diagnosis of gout were enrolled equally in 1 of 2 treatment groups, once a day placebo or febuxostat 40 mg or 80 mg based on serum urate levels.
Period: Overall Study
Arm/Group | Febuxostat 40 mg or 80 mg | Placebo
Started | 157 | 157
Completed | 93 | 90
Not Completed | 64 | 67
Not completed — Adverse Event | 10 | 6
Not completed — Major Protocol Deviation | 2 | 0
Not completed — Lost to Follow-up | 23 | 23
Not completed — Voluntary Withdrawal | 20 | 36
Not completed — Other | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat 40 mg or 80 mg | Placebo | Total
Number analyzed (Participants) | 157 | 157 | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (12.36) | 50.1 (11.72) | 50.8 (12.04)
Age, Customized [Number; unit: participants]
  <45 years | 49 | 42 | 91
  45 to <65 years | 85 | 99 | 184
  ≥65 years | 23 | 16 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 143 | 145 | 288
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 8 | 10 | 18
  Black or African American | 25 | 24 | 49
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 119 | 121 | 240
  Other | 3 | 2 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 26 | 36 | 62
  Not Hispanic or Latino | 131 | 121 | 252
Region of Enrollment [Number; unit: participants]
  United States | 157 | 157 | 314
Height [Mean (Standard Deviation); unit: cm] | 176.3 (9.22) | 176.5 (8.36) | 176.4 (8.79)
Weight [Mean (Standard Deviation); unit: kg] | 102.8 (20.88) | 100.7 (21.20) | 101.7 (21.04)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.1 (6.40) | 32.3 (6.23) | 32.7 (6.32)
BMI Categories [Number; unit: participants]
  <25 kg/m^2 | 11 | 11 | 22
  25 to <30 kg/m^2 | 37 | 46 | 83
  ≥30 kg/m^2 | 109 | 100 | 209
Smoking History [Number; unit: participants]
  Never Smoked | 84 | 94 | 178
  Current Smoker | 32 | 25 | 57
  Ex-Smoker | 41 | 38 | 79
Alcohol History [Number; unit: participants]
  Never Drank | 37 | 35 | 72
  Current Drinker | 103 | 106 | 209
  Ex-Drinker | 17 | 16 | 33
Renal History (Modification of Diet in Renal Disease [MDRD]) [Number; unit: participants]
  Moderately Impaired MDRD | 3 | 2 | 5
  Mildly Impaired MDRD | 105 | 115 | 220
  Normal MDRD | 49 | 40 | 89

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Month 24 in the Modified Sharp/Van Der Heijde Erosion Score of the Single Affected Joint
Description: The single affected joint was defined as the joint with the history of the first acute gout flare. Radiographs (X-rays) of this single joint in the hands or feet were evaluated using the modified Sharp/van der Heijde method. Each erosion was assessed using a 4-point scale where 0=no erosions (best) to 3=large erosion passing the mid-line (worst). Individual erosion scores were summed to a maximum erosion score of 5 for joints in the hands and 10 for joints in the feet. Higher scores indicated more joint damage. A negative change from Baseline indicated improvement.
Time Frame: Baseline and Month 24
Population: Full Analysis Set included all randomized participants who received at least one dose of study medication. Participants were analyzed according to the treatment group to which they actually received. Participants with data available for analysis and missing values at Month 24 imputed using linear extrapolation are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Febuxostat 40 mg or 80 mg | Placebo
Number analyzed (Participants) | 86 | 82
score on a scale
  Baseline | 0.16 (0.444) | 0.11 (0.438)
  Change from Baseline at Month 24 | 0.01 (0.330) | 0.01 (0.248)
Statistical Analysis 1: Comparison: Febuxostat 40 mg or 80 mg vs Placebo; Change from Baseline at Month 24; Test type: Superiority or Other; p = 0.472, Ranked Analysis of Covariance (ANCOVA); Baseline modified Sharp/van der Heijde Erosion Score as a covariate

2. Secondary Outcome: Mean Change From Baseline to Month 24 in the Modified Sharp/Van Der Heijde Total Scores From Full Hands and Feet Radiographs
Description: Radiographs (X-rays) of 40 joints in the hands and 12 joints in the feet were evaluated using the modified Sharp/van der Heijde method. Each erosion was assessed using a 4-point scale where 0=no erosions (best) to 3=large erosion passing the mid-line (worst) for a total erosion score range of 0 to 320. Joint space narrowing (JSN) was assessed using a 5-point scale where 0=normal (best) to 4=absence of joint space, presumptive evidence of ankyloses, or complete luxation (worst) for a total JSN score range of 0 to 208. The Erosion Score and the JSN Score were combined for a total possible score of 0 to 528. Higher scores indicated more joint damage. A negative change from Baseline indicated improvement.
Time Frame: Baseline and Month 24
Population: Full Analysis Set included all randomized participants who received at least one dose of study medication. Participants were analyzed according to the treatment group to which they actually received. Participants with data available at Baseline and Month 24 are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Febuxostat 40 mg or 80 mg | Placebo
Number analyzed (Participants) | 91 | 86
score on a scale
  Baseline | 4.98 (9.707) | 4.56 (8.631)
  Change from Baseline at Month 24 (n=78,74) | 0.31 (2.447) | 0.29 (1.746)
Statistical Analysis 1: Comparison: Febuxostat 40 mg or 80 mg vs Placebo; Change from Baseline at Month 24; Test type: Superiority or Other; p = 0.548, Ranked ANCOVA; Baseline modified Sharp/van der Heijde Total Score from full hands and feet as a covariate

3. Secondary Outcome: Mean Change From Baseline to Month 24 in the Modified Sharp/Van Der Heijde Erosion Scores From Full Hands and Feet Radiographs
Description: Radiographs (X-rays) of 40 joints in the hands and 12 joints in the feet were evaluated using the modified Sharp/van der Heijde method. Each erosion was assessed using a 4-point scale where 0=no erosions (best) to 3=large erosion passing the mid-line (worst) for a total erosion score range of 0 to 320. Higher scores indicated more joint damage. A negative change from Baseline indicated improvement.
Time Frame: Baseline and Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Febuxostat 40 mg or 80 mg | Placebo
Number analyzed (Participants) | 91 | 86
score on a scale
  Baseline | 0.36 (1.160) | 0.17 (0.473)
  Change from Baseline at Month 24 (n=78,74) | 0.17 (1.709) | 0.11 (0.969)
Statistical Analysis 1: Comparison: Febuxostat 40 mg or 80 mg vs Placebo; Change from Baseline at Month 24; Test type: Superiority or Other; p = 0.389, Ranked ANCOVA; Baseline modified Sharp/van der Heijde Erosion Score from full hands and feet as a covariate

4. Secondary Outcome: Mean Change From Baseline to Month 24 in the Rheumatoid Arthritis MRI Scoring System (RAMRIS) Score of the Single Affected Joint
Description: The single affected joint was defined as the joint with the history of the first acute gout flare. Magnetic Resonance Imaging (MRI) was evaluated using the Rheumatoid Arthritis MRI Score (RAMRIS). Bone erosion in the proximal and distal location were each assessed in the affected joint using an 11-point scale where 0=no erosion (best) to 10=91-100% bone eroded (worst) for a bone erosion score range of 0 to 20. Bone marrow edema in the proximal and distal location were each assessed using a 4-point scale where 0=no edema (best) to 3=67-100% edema (worst) for a bone marrow edema (BME) score range of 0 to 6. Synovitis was assessed in the affected joint using a 4-point scale where 0=normal (best) to 3=severe (worst). Higher scores indicated more joint damage. A negative change from Baseline indicated improvement.
Time Frame: Baseline and Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Febuxostat 40 mg or 80 mg | Placebo
Number analyzed (Participants) | 157 | 157
score on a scale
  Synovitis:Baseline (BL)(n=82,76) | 1.29 (0.782) | 1.09 (0.687)
  Synovitis:Change from Baseline (n=75,67) | -0.43 (0.713) | -0.07 (0.531)
  Erosion (Distal+Proximal):Baseline (n=84,77) | 1.63 (0.935) | 1.48 (0.916)
  Erosion (Distal+Proximal):Change from BL(n=79,69) | -0.01 (0.702) | 0.04 (0.475)
  Edema (Distal+Proximal):Baseline (BL) (n=81,75) | 0.73 (1.022) | 0.51 (0.919)
  Edema (Distal+Proximal):Change from BL(n=77,66) | -0.36 (0.916) | -0.10 (0.962)
Statistical Analysis 1: Comparison: Febuxostat 40 mg or 80 mg vs Placebo; Synovitis: Change from Baseline at Month 24; Test type: Superiority or Other; p < 0.001, Ranked ANCOVA; Baseline RAMRIS Synovitis Score as a covariate
Statistical Analysis 2: Comparison: Febuxostat 40 mg or 80 mg vs Placebo; Erosion(Distal+Proximal): Change from Baseline at Month 24; Test type: Superiority or Other; p = 0.634, Ranked ANCOVA; Baseline RAMRIS Erosion(Distal+Proximal) Score as a covariate
Statistical Analysis 3: Comparison: Febuxostat 40 mg or 80 mg vs Placebo; Edema(Distal+Proximal): Change from Baseline at Month 24; Test type: Superiority or Other; p = 0.307, Ranked ANCOVA; Baseline RAMRIS Edema(Distal+Proximal) Score as a covariate

5. Secondary Outcome: Mean Change From Baseline to Month 24 in the Modified Sharp/Van Der Heijde Total Score of the Single Affected Joint
Description: The single affected joint was defined as the joint with the history of the first acute gout flare. Radiographs (X-rays) of the single affected joint in the hands or feet were evaluated using the modified Sharp/van der Heijde method. Each erosion was assessed using a 4-point scale where 0=no erosions (best) to 3=large erosion passing the mid-line (worst) and Joint space narrowing (JSN) was assessed using a 5-point scale where 0=normal (best) to 4=absence of joint space, presumptive evidence of ankyloses, or complete luxation (worst). The Erosion Score and the JSN Score were summed for the Total Score. Higher scores indicated more joint damage. A negative change from Baseline indicated improvement.
Time Frame: Baseline and Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Febuxostat 40 mg or 80 mg | Placebo
Number analyzed (Participants) | 86 | 82
score on a scale
  Baseline | 0.85 (1.057) | 0.77 (1.022)
  Change from Baseline at Month 24(n=81,76) | 0.00 (0.602) | 0.05 (0.361)
Statistical Analysis 1: Comparison: Febuxostat 40 mg or 80 mg vs Placebo; Change from Baseline at Month 24; Test type: Superiority or Other; p = 0.122, Ranked ANCOVA; Baseline modified Sharp/van der Heijde Total Score as a covariate

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events, regardless of relationship to study drug, that started on or after the first dose of study drug and no more than 30 days after last dose of study drug (Up to 25 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Febuxostat 40 mg or 80 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 13/157 | 11/157
Other Adverse Events (participants affected / at risk) | 73/157 | 67/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 40 mg or 80 mg (N=157) | Placebo (N=157)
Cardiac failure congestive (Cardiac disorders) | 1 | 1 — One treatment-emergent death occurred during treatment with febuxostat and is not related.
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1 — One treatment-emergent death occurred during treatment with placebo and is not related.
Vitreous haemorrhage (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Hepatic infection (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Chest wall abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 40 mg or 80 mg (N=157) | Placebo (N=157)
Diarrhoea (Gastrointestinal disorders) | 9 | 6
Oedema peripheral (General disorders) | 8 | 5
Upper respiratory tract infection (Infections and infestations) | 15 | 16
Aspartate aminotransferase increased (Investigations) | 11 | 6
Blood creatine phosphokinase increased (Investigations) | 9 | 11
Alanine aminotransferase increased (Investigations) | 10 | 6
Gamma-glutamyltransferase increased (Investigations) | 6 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 8
Headache (Nervous system disorders) | 5 | 10
Hypertension (Vascular disorders) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.